CLINICAL TRIAL: NCT01237041
Title: Free Fatty Acids, Body Weight, and Growth Hormone Secretion in Children
Brief Title: Free Fatty Acids, Body Weight, and Growth Hormones Secretion in Children
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study Medication unavailable
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jack Yanovski, M.D., Chief, Section on Growth and Obesity, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 110004; 11-CH-0004 (Other: NIH Clinical Center Protocol Number)
Record Dates: First submitted 2010-11-06; First posted 2010-11-09 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Obesity; Short Stature; Growth Hormone Deficiency
Keywords: Child; Body Fat; Niacin; Growth Hormone; Obesity; Overweight; Growth Hormones; Short Stature; Children
MeSH Terms: conditions — Obesity; Dwarfism; Dwarfism, Pituitary; Overweight

STUDY DESIGN:
Intervention Model Description: First, we conducted dose-establishing studies using 250mg every 2 hours x 3 doses (2 subjects), 500mg every two hours x 3 doses (5 subjects), and 500mg hourly x 4 doses (5 subjects). This dose-establishing study was followed by the randomized crossover trial using 500mg hourly x 4 doses in conjunction with growth hormone stimulation testing. The RCT was terminated early because of inability to obtain necessary study medications.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking only during the two arms of the randomized trial portion of the study, not during the dose-finding arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Niacin First (Experimental): Subjects receive niacin 500mg hourly for 4 hours on day 1 (at 7:30am, 8:30am, 9:30am, and 10:30am) then cross over to receive placebo hourly for 4 hours on day 2 at (7:30am, 8:30am, 9:30am, and 10:30am).
  Interventions: Drug: Niacin First; Drug: Placebo First
- Placebo First (Experimental): Subjects receive placebo hourly for 4 hours on day 1 (at 7:30am, 8:30am, 9:30am, and 10:30am) then cross over to receive niacin hourly for 4 hours on day 2 (at 7:30am, 8:30am, 9:30am, and 10:30am).
  Interventions: Drug: Niacin First; Drug: Placebo First
- Dose-Establishing Study 1 Niacin 250mg (Experimental): Subjects received Niacin 250 mg every 2 hours for 3 doses (at 6am, 8am, and 10am).
  Interventions: Drug: Dose-Establishing Study 1 Niacin 250mg
- Dose-Establishing Study 1 Niacin 500mg (Experimental): Subjects received Niacin 500 mg every 2 hours for 3 doses (at 6am, 8am, and 10am).
  Interventions: Drug: Dose-Establishing Study 1 Niacin 500mg
- Dose-Establishing Study 2 Niacin 500mg (Experimental): Subjects received Niacin 500 mg hourly for 4 doses (administered at 7:30am, 8:30am, 9:30am, and 10:30am).
  Interventions: Drug: Dose-Establishing Study 2 Niacin 500mg

INTERVENTIONS:
Drug: Niacin First — Niacin 500 mg po four times on one of the inpatient days, then placebo on another inpatient day
  Other Names: RCT Niacin First
  Arms: Niacin First; Placebo First
Drug: Placebo First — Placebo po four times on one of the inpatient days, then Niacin 500 mg po four times on another inpatient day
  Other Names: RCT Placebo First
  Arms: Niacin First; Placebo First
Drug: Dose-Establishing Study 1 Niacin 250mg — Niacin 250 mg po three times at 2 hour intervals on an inpatient day
  Other Names: Open-Label Niacin 250mg x 3 doses
  Arms: Dose-Establishing Study 1 Niacin 250mg
Drug: Dose-Establishing Study 1 Niacin 500mg — Niacin 500 mg po three times at 2 hour intervals on an inpatient day
  Other Names: Open-Label Niacin 500mg x 3 doses
  Arms: Dose-Establishing Study 1 Niacin 500mg
Drug: Dose-Establishing Study 2 Niacin 500mg — Open-Label Niacin 500mg four times at 1 hour intervals on an inpatient day
  Other Names: Open-Label Niacin 500mg x four doses
  Arms: Dose-Establishing Study 2 Niacin 500mg

SUMMARY:
Background:

- Overweight and obese children and adults often have lower levels of growth hormone in the blood. Regulation of growth hormone may be tied to weight and free fatty acids in the blood. Current tests of growth hormone (such as those used when evaluating the heights of children who are markedly shorter than other children of comparable age) may be affected by other factors, including obesity. Researchers are interested in evaluating the levels of growth hormone and free fatty acids in the blood of children between 7 and 14 years of age who weigh more than children of a comparable age, or who are shorter than other children of a comparable age and have been recommended for growth hormone testing as part of an evaluation for their height.

Objectives:

- To determine the effect of changes in free fatty acids in the blood on changes in growth hormone secretion in overweight or shorter children and young adolescents.

Eligibility:

- Children and adolescents between 7 and 14 years of age who weigh more than or are shorter than other children of a comparable age and do not have any medical illnesses.

Design:

* Participants will have two study visits, one of which will be a half day screening visit in the outpatient clinic and one of which will require 2 nights as an inpatient at the National Institutes of Health Clinical Center.
* Participants should not eat or drink anything except water after 10 PM the night before or on the morning of the screening visit.
* At the screening visit, participants will have a physical examination and medical history, provide blood and urine samples, have an oral glucose tolerance test (to check blood sugar levels), and have an x-ray of the left hand to check bone age.
* The inpatient study visit will involve a physical examination and medical history, a full x-ray scan to study body fat and muscle, frequent blood tests throughout the visit, and various medications to stimulate growth hormone production and lower levels of free fatty acids in the blood.

DETAILED DESCRIPTION:
Obese children and adults display lower spontaneous and stimulated growth hormone (GH) secretion. It is presumed that dysregulation of some of the factors normally involved in controlling GH secretion underlies the hyposomatotropinemia of obesity, given that GH production usually normalizes after weight loss. Free fatty acids (FFA) are one factor thought to be involved in regulation of GH secretion. Niacin is a nicotinic acid derivative that inhibits lipolysis and lowers circulating FFA concentrations. Nicotinic acid derivatives have been used in several adult studies examining GH secretion. Specifically in obese adults, inhibition of lipolysis has been found to increase spontaneous and stimulated GH production, presumably due to direct effects of FFA on hypothalamic GH-regulating neurons. Thus far no pediatric studies have examined the effects of niacin on GH secretion, and there is only one small pediatric study of normal weight prepubertal children growing at the 5th-10th percentile in height has tested the effects of lipolytic inhibition by acipimox (a related medication also derived from nicotinic acid) on GH secretion. There are no data in obese children demonstrating the effects of inhibition of lipolysis on GH secretion.

We propose to investigate one of the mechanisms through which high adiposity alters GH secretion in children by testing the effects of inhibiting lipolysis. First we will conduct dose establishing studies to determine the appropriate dose of niacin needed to suppress FFA concentrations in children. We will then conduct the main study, designed as a pilot randomized, double-blind placebo controlled trial of niacin administration, to assess its effects on stimulated GH secretion. We hypothesize that in overweight children niacin will lead to a fall in free fatty acid concentrations and consequently a rise in stimulated GH secretion. We further hypothesize that the overweight subjects will demonstrate stimulated GH secretion profiles with niacin similar to those of control subjects who receive placebo. We expect this pilot study may help improve how diagnostic testing is carried out for growth hormone deficiency in children.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will qualify for the overweight group for the dose-establishing studies 1 and 2 and main study) if they meet the following criteria:

1. Good general health.
2. Age greater than or equal to 7 and less than 15 years.
3. Tanner stage I, II or III for the breast among girls and testes less than10 mL for boys based upon an examination by a trained physician or nurse practitioner.
4. Weight > 30 kg.
5. Fasting plasma glucose < 100 mg/dL, 2 hour post-dextrose glucose < 140 mg/dL, and HgbA1C less than or equal to 6.4%.
6. Females who are age 10 or greater must have a negative pregnancy test.
7. Body mass index greater than or eqaul to 95th percentile determined by Centers for Disease Control age and sex specific data (given that most pathology of obesity does not usually emerge until children cross the 95th percentile).
8. No evidence of growth failure as defined as height > 5th percentile.

Subjects will qualify for the non-overweight control group (for the main study only) if they meet the following criteria:

1. Recommended by a pediatric endocrinologist to undergo GH stimulation testing to establish the diagnosis of GH-deficiency.
2. Good general health.
3. Age greater than or equal to 7 and less than15 years.
4. Tanner stage I, II or III for the breast among girls and testes less than 10 mL for boys based upon an examination by a trained physician or nurse practitioner.
5. Weight > 30 kg.
6. Fasting plasma glucose < 100 mg/dL, 2 hour post-dextrose glucose < 140 mg/dL, and HgbA1C less than or equal to 6.4%.
7. Females who are age 10 or greater must have a negative pregnancy test.
8. Height < 5th percentile.
9. BMI between the 5th and 85th percentiles determined by Centers for Disease Control age and sex specific data.
10. Birth weight and length not consistent with small for gestational age (SGA) criteria or a history of intrauterine growth restriction (IUGR) based on recall history.

EXCLUSION CRITERIA (for the dose-establishing sutides 1 and 2, and the main study):

Subjects will be excluded if they have any of the following:

1. Baseline creatinine greater than or equal to 1.0 mg/dl.
2. Significant cardiac or pulmonary disease likely to or resulting in hypoxia or decreased perfusion.
3. Hepatic disease with elevated liver function tests (ALT or AST)greater than or equal to 1.5 the upper limits of normal.
4. Pregnancy.
5. Evidence for impaired glucose tolerance or Type 2 diabetes, including fasting plasma glucose greater than or equal to 100 mg/dL, 2 hour post-dextrose glucose greater than or equal to 140 mg/dL, or HgbA1C > 6.4%.
6. Presence of other endocrinologic disorders leading to obesity (e.g. Cushing Syndrome).
7. Any disorder that is known to affect GH secretion (e.g. untreated hypothyroidism) or use of any medication known to affect GH levels (including glucocorticoids and GH itself).
8. Any other disorder that is known to affect stature including skeletal dysplasias.
9. Recent use (within two years) of anorexiant medications, stimulant medications, or other medications felt to impact growth.
10. Individuals who have, or whose parent or guardians have, current substance abuse or a psychiatric disorder or other condition that, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study.
11. Individuals receiving medical treatment other than diet for hypertension or dyslipidemia.
12. Individuals with evidence of precocious puberty as defined as palpable breast tissue noted in females before the age of 7, testicular size greater than or equal to 4cc in males before the age of 9, or bone age advancement more than 2 SD for chronologic age.
13. Individuals receiving androgen or estrogen hormone therapy.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Tauber M, Moulin P, Pienkowski C, Jouret B, Rochiccioli P. Growth hormone (GH) retesting and auxological data in 131 GH-deficient patients after completion of treatment. J Clin Endocrinol Metab. 1997 Feb;82(2):352-6. doi: 10.1210/jcem.82.2.3726. PMID 9024217
- [Background] Cohen P, Rogol AD, Deal CL, Saenger P, Reiter EO, Ross JL, Chernausek SD, Savage MO, Wit JM; 2007 ISS Consensus Workshop participants. Consensus statement on the diagnosis and treatment of children with idiopathic short stature: a summary of the Growth Hormone Research Society, the Lawson Wilkins Pediatric Endocrine Society, and the European Society for Paediatric Endocrinology Workshop. J Clin Endocrinol Metab. 2008 Nov;93(11):4210-7. doi: 10.1210/jc.2008-0509. Epub 2008 Sep 9. PMID 18782877
- [Background] Zucchini S, Pirazzoli P, Baronio F, Gennari M, Bal MO, Balsamo A, Gualandi S, Cicognani A. Effect on adult height of pubertal growth hormone retesting and withdrawal of therapy in patients with previously diagnosed growth hormone deficiency. J Clin Endocrinol Metab. 2006 Nov;91(11):4271-6. doi: 10.1210/jc.2006-0383. Epub 2006 Aug 15. PMID 16912138
- [Background] Galescu OA, Crocker MK, Altschul AM, Marwitz SE, Brady SM, Yanovski JA. A pilot study of the effects of niacin administration on free fatty acid and growth hormone concentrations in children with obesity. Pediatr Obes. 2018 Jan;13(1):30-37. doi: 10.1111/ijpo.12184. Epub 2016 Sep 21. PMID 27654882

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 37 enrolled, two withdrew from the study before being studied. 16 were ineligible. 7 subjects completed the first niacin dose-establishing protocol. 5 completed the second phase pilot study. A total of 5 subjects were randomized in the main study. Two subjects were eligible, but were never studied due to unavailability of study medications.
Groups:
- Niacin First: Subjects receive niacin on day 1 then cross over to receive placebo on day 2.
  Niacin: 500 mg po four times on one of the inpatient day
  Placebo po four times on the next inpatient day
- Placebo First: Subjects receive placebo on day 1 then cross over to receive niacin on day 2
  Placebo po four times on an inpatient day Niacin: 500 mg po four times on the next inpatient day
Period: Overall Study
Arm/Group | Niacin First | Placebo First | Dose-Establishing Study 1 Niacin 250mg | Dose-Establishing Study 1 Niacin 500mg | Dose-Establishing Study 2 Niacin 500mg
Started | 2 | 3 | 2 | 5 | 5
Completed | 2 | 3 | 2 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Niacin First: Subjects receive niacin on day 1 then cross over to receive placebo on day 2.
  Niacin: 500 mg po four times on one of the inpatient days
  Placebo
- Placebo First: Subjects receive placebo on day 1 then cross over to receive niacin on day 2
  Niacin: 500 mg po four times on one of the inpatient days
  Placebo
- Dose-Establishing Study 1 Niacin 250mg: Niacin 250mg x 3 doses 2 hours apart at 6AM, 8AM, and 10AM
- Dose-Establishing Study 1 Niacin 500mg: Niacin 500mg x 3 doses 2 hours apart 6AM, 8AM, and 10AM
- Dose-Establishing Study 2 Niacin 500mg: Niacin 500mg x 4 doses 1 hours apart 7:30AM, 8:30AM, 9:30AM, and 10:30AM
- Total: Total of all reporting groups
Arm/Group | Niacin First | Placebo First | Dose-Establishing Study 1 Niacin 250mg | Dose-Establishing Study 1 Niacin 500mg | Dose-Establishing Study 2 Niacin 500mg | Total
Number analyzed (Participants) | 2 | 3 | 2 | 5 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (2.3) | 10.8 (1.3) | 10.5 (2.2) | 9.7 (2.0) | 9.3 (1.9) | 10.1 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 3 | 1 | 5
  Male | 2 | 2 | 2 | 2 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 3 | 2 | 5 | 5 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 3 | 2 | 7
  White | 2 | 2 | 0 | 2 | 3 | 9
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 2 | 5 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Growth Hormone Secretion Area Under the Curve in Response to Niacin and Placebo Over Time
Description: Growth hormone Area Under the Curve in response to niacin versus placebo over 4 hours. For growth hormone, samples collected at 0, 30, 60, 90, 120, 150, 180, 210, and 240 minutes.
Time Frame: 4 hours
Population: No placebo was given during the dose-establishing arms, so no data are reported for placebo.
Measure: Mean (Standard Deviation); unit: min*ng/mL
Groups:
- All Randomized Subjects: Results of both randomization orders to assess effect of niacin
- Dose-Establishing Study 1 Niacin 250mg: Dose-Establishing Study 1 Niacin 250mg every 2 hours for 3 doses
- Dose-Establishing Study 1 Niacin 500mg: Dose-Establishing Study 1 Niacin 500mg every 2 hours for 3 doses
- Dose-Establishing Study 2 Niacin 500mg: Dose-Establishing Study 2 Niacin 500mg every 1 hour for 4 doses
Arm/Group | All Randomized Subjects | Dose-Establishing Study 1 Niacin 250mg | Dose-Establishing Study 1 Niacin 500mg | Dose-Establishing Study 2 Niacin 500mg
Number analyzed (Participants) | 5 | 2 | 5 | 5
min*ng/mL
  Niacin | 589.6 (437.6) | 32.0 (20.7) | 84.0 (68.6) | 394.6 (217.9)
  Placebo: number analyzed (Participants) | 5 | 0 | 0 | 0
  Placebo | 638.5 (513.9) |  |  |
Statistical Analysis 1: Comparison: Dose-Establishing Study 1 Niacin 250mg vs Dose-Establishing Study 1 Niacin 500mg vs Dose-Establishing Study 2 Niacin 500mg; ANOVA to compare AUC of GH among groups; Test type: Superiority — Univariate ANOVA; p = .016, ANOVA — A priori threshold p<0.05; Comparison of 3 dose-finding groups. Post-hoc comparisons between groups also done

2. Secondary Outcome: Free Fatty Acids (FFA) Area Under the Curve in Response to Niacin and Placebo Over 4 Hours
Description: Effect of niacin vs placebo on Free Fatty Acids (FFA) Area Under the Curve in response to Niacin and Placebo over 4 hours. For FFA, samples collected at 0, 30, 60, 90, 120, 150, 180, 210, and 240 minutes
Time Frame: 4 hours
Population: Dose-establishing participants did not have placebo, so there are no data for those cells.
Measure: Mean (Standard Deviation); unit: Min*UEq/L
Arm/Group | All Randomized Subjects | Dose-Establishing Study 1 Niacin 250mg | Dose-Establishing Study 1 Niacin 500mg | Dose-Establishing Study 2 Niacin 500mg
Number analyzed (Participants) | 5 | 2 | 5 | 5
Min*UEq/L
  Niacin FFA AUC | 37567 (12065) | 164056 (110047) | 94346 (42439) | 48870 (20243)
  Placebo FFA AUC: number analyzed (Participants) | 5 | 0 | 0 | 0
  Placebo FFA AUC | 106047 (37010) |  |  |
Statistical Analysis 1: Comparison: Dose-Establishing Study 1 Niacin 250mg vs Dose-Establishing Study 1 Niacin 500mg vs Dose-Establishing Study 2 Niacin 500mg; Analysis of FFA Area Under Curve in dose-finding studies. Data were log-transformed before analysis; Test type: Superiority — ANOVA of the 3 dose-finding groups. Data transformed using log(10) for analysis; p = .043, ANOVA — A priori threshold for significance p<0.05

3. Secondary Outcome: Growth Hormone-releasing Hormone (GHRH) Area Under the Curve in Response to Niacin and Placebo Over 4 Hours
Description: Growth hormone-releasing hormone (GHRH) Area Under the Curve in response to Niacin and Placebo over 4 hours. For GHRH, samples collected at 0, 60, 120, 180, and 240 minutes.
Time Frame: 4 hours
Population: Dose-establishing participants did not have placebo, so there are no data for those cells.
Measure: Mean (Standard Deviation); unit: min*pg/mL
Arm/Group | All Randomized Subjects | Dose-Establishing Study 1 Niacin 250mg | Dose-Establishing Study 1 Niacin 500mg | Dose-Establishing Study 2 Niacin 500mg
Number analyzed (Participants) | 5 | 2 | 5 | 5
min*pg/mL
  Niacin GHRH | 2535 (898.2) | 2415 (129.9) | 2548 (637.5) | 5382 (8090.1)
  Placbo GHRH: number analyzed (Participants) | 5 | 0 | 0 | 0
  Placbo GHRH | 2283 (1505.6) |  |  |
Statistical Analysis 1: Comparison: Dose-Establishing Study 1 Niacin 250mg vs Dose-Establishing Study 1 Niacin 500mg vs Dose-Establishing Study 2 Niacin 500mg; ANOVA, 3 dose-finding groups; Test type: Superiority; p = 0.543, ANOVA

4. Secondary Outcome: Somatostatin (SST) Area Under the Curve in Response to Niacin and Placebo Over 4 Hours
Description: Effect of niacin vs placebo on Somatostatin (SST) Area Under the Curve in response to Niacin and Placebo over 4 hours. For somatostatin, samples collected at 0, 60, 120, 180, and 240 minutes.
Time Frame: 4 hours
Population: Dose-establishing participants did not have placebo, so there are no data for those cells. Dose-establishing study 1 niacin 250mg participants did not have somatostatin measured, so those cells are also not completed
Measure: Mean (Standard Deviation); unit: min*pg/mL
Arm/Group | All Randomized Subjects | Dose-Establishing Study 1 Niacin 250mg | Dose-Establishing Study 1 Niacin 500mg | Dose-Establishing Study 2 Niacin 500mg
Number analyzed (Participants) | 5 | 0 | 5 | 5
min*pg/mL
  Niacin Somatostatin | 1329 (615.7) |  | 849.8 (484.5) | 1578 (692.1)
  Placebo Somatostatin: number analyzed (Participants) | 5 | 0 | 0 | 0
  Placebo Somatostatin | 1248 (461.5) |  |  |
Statistical Analysis 1: Comparison: Dose-Establishing Study 1 Niacin 500mg vs Dose-Establishing Study 2 Niacin 500mg; ANOVA, 2 groups, essentially an unpaired t-test; Test type: Superiority; p = .113, ANOVA

ADVERSE EVENTS:
Time Frame: 4 hours
Description: Adverse events by hourly questionnaire
Groups:
- All Randomized Subjects: Results of both randomization orders to assess effect of Niacin 500mg every 1 hour for 4 doses
- Dose-Finding Study 1 Niacin 250mg: Results from Niacin 250mg every 2 hours for 3 doses
- Dose-Finding Study 1 Niacin 500mg: Results from Niacin 500mg every 2 hours for 3 doses
- Dose-Finding Study 2 Niacin 500mg: Results from Niacin 500mg every 1 hour for 4 doses
Arm/Group | All Randomized Subjects | Dose-Finding Study 1 Niacin 250mg | Dose-Finding Study 1 Niacin 500mg | Dose-Finding Study 2 Niacin 500mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/5 | 0/2 | 1/5 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Randomized Subjects (N=5) | Dose-Finding Study 1 Niacin 250mg (N=2) | Dose-Finding Study 1 Niacin 500mg (N=5) | Dose-Finding Study 2 Niacin 500mg (N=5)
Nausea (Gastrointestinal disorders) | 3 (8) | 0 (0) | 1 (3) | 3 (9) — Nausea during niacin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT01237041/Prot_SAP_000.pdf